CLINICAL TRIAL: NCT04524754
Title: Prevalence and Outcomes of Olfactory and Gustatory Dysfunctions in Patients With COVID-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed Shehata Taha, Professor Doctor, Ain Shams University
Other Study IDs: FMASUP46a/2020
Record Dates: First submitted 2020-08-21; First posted 2020-08-24 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Anosmia
MeSH Terms: conditions — Anosmia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prevalence and Outcomes of Olfactory and Gustatory Dysfunctions in Patients with COVID-19

DETAILED DESCRIPTION:
AIM OF THE STUDY AND WORK PLAN COVID-19 Hospitalized patients with confirmed diagnosis of disease will

1. undergo questionnaire for prevalence of Anosmia/dysgeusia
2. linking the anosmia/dysgeusia to the degree of disease and treatment outcomes.
3. looking to improvement in anosmia/dysgeusia and its timing,

METHODOLOGY Ethical committee approval for the current study protocol will be obtained. Patients will be invited to participate and the informed consent will be signed.

Subjects and Setting:

The clinical data of 218 patients with laboratory-confirmed COVID-19 infection will be collected from Ain Shams University Hospitals. In addition, other patients, infected physicians and nurses may voluntarily enroll in the study. Comorbidities as diabetes mellitus or hypertension, and chronic treatment lines taken will be documented, and considered in the analysis of the data. Patients would be receiving the ASU treatment protocol for covid 19.

The following inclusion criteria will be considered: adult (>18 year); laboratory-confirmed COVID-19 infection (reverse transcription polymerase chain reaction, RT-PCR). The following exclusion criteria will be considered: patients with olfactory or gustatory dysfunctions before the epidemic; patients without a laboratory-confirmed COVID-19 infection diagnosis; patients who were in the intensive care unit at the time of the study (due to their health status).

Clinical Outcomes Clinical data will be collected during the ear, nose, and throat (ENT) consultation; in the patient's room.

Questions about olfactory function; questions investigating gustatory function; and questions about the treatment of the COVID-19 infection. All patients will be asked to answer these questions.

Olfactory and Gustatory Outcomes The occurrence of olfactory dysfunction has been identified through several questions including social, eating, annoyance, and anxiety questions. The rest of the olfactory and gustatory questions will be based on the smell and taste. The questions have been chosen to characterize the variation, timing and associated-symptoms of both olfactory and gustatory dysfunctions, and, therefore, they suggest a potential etiology. Also the mean recovery time of olfaction will be assessed through 4 defined propositions: 1-4 days; 5-8 days; 9-14 days and >15 days.

Statistical Analysis First, the following descriptive analysis will be done: frequency, percentages, mean and standard deviation (SD). Thereafter, a comparison will be done using Student t-test for quantitative variables and Fisher exact test for qualitative variables.

Statistical Package Data entry and statistical analysis will be done using Statistical Package for Social Science (SPSS) version 20.0.

ELIGIBILITY:
Inclusion Criteria:

* adult (>18 year); laboratory-confirmed COVID-19 infection (reverse transcription polymerase chain reaction, RT-PCR).

Exclusion Criteria:

* patients with olfactory or gustatory dysfunctions before the epidemic; patients without a laboratory-confirmed COVID-19 infection diagnosis; patients who were in the intensive care unit at the time of the study (due to their health status).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 218 patients with laboratory-confirmed COVID-19 infection will be collected from Ain Shams University Hospitals
Sampling Method: Non-Probability Sample
Enrollment: 218 (Estimated)
Dates: Start 2020-07-11 (Actual); Primary Completion 2020-09-11 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
olfaction | one month
  subjective on a scale from 1 to 5 ( 1 is the least and 5 is the best ) , the score will be recorded for olfaction before and after the olfactory loss

SECONDARY OUTCOMES:
gustation | one month
  subjective on a scale from 1 to 5 ( 1 is the least and 5 is the best ) , , the score will be recorded for gustation before and after the gustatory loss

CONTACTS AND LOCATIONS:
Overall Officials: ethical committee, Study Director — Ain Shams University
Locations (1):
- Ain shams Univesrity, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Moein ST, Hashemian SM, Mansourafshar B, Khorram-Tousi A, Tabarsi P, Doty RL. Smell dysfunction: a biomarker for COVID-19. Int Forum Allergy Rhinol. 2020 Aug;10(8):944-950. doi: 10.1002/alr.22587. Epub 2020 Jun 18. PMID 32301284
- [Background] Spinato G, Fabbris C, Polesel J, Cazzador D, Borsetto D, Hopkins C, Boscolo-Rizzo P. Alterations in Smell or Taste in Mildly Symptomatic Outpatients With SARS-CoV-2 Infection. JAMA. 2020 May 26;323(20):2089-2090. doi: 10.1001/jama.2020.6771. PMID 32320008